CLINICAL TRIAL: NCT04086251
Title: Remote Electronic Patient Monitoring in Oncology Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Gaido Health (Industry)
Collaborators: The Guthrie Clinic (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: GHBC-0719
Record Dates: First submitted 2019-07-22; First posted 2019-09-11 (Actual); Last update posted 2019-09-11 (Actual); Status verified 2019-09

CONDITIONS: Cancer
Keywords: Neoplasm; Malignancy; Oncology; Remote patient monitoring
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Gaido Intervention (Experimental): All patients enrolled in the study will participate in the Gaido Intervention, which entails wearing the Biovotion Everion continuously and take blood pressure and oral temperature spot checks per clinician orders. Patients will also be responsible for filling out PRO surveys and any surveys that trigger as a result of their vital signs falling outside of tailored thresholds.
  Interventions: Other: Gaido

INTERVENTIONS:
Other: Gaido — Patients will participate for up to 21 days. Over the course of the study, 25-100 patients will be enrolled.
  Other Names: Remote electronic patient monitoring

SUMMARY:
The goal of this research is to study an intervention, which the investigators call "Remote Electronic Patient Monitoring," that entails vital sign data (enabled with smart algorithms for notification) and patient-reported outcomes (PROs), (such as physical and psychological symptoms) intended to address and manage any concerning issues and or diagnoses identified.

Specifically, the plan is a study of oncology patients who will use the Gaido system for up to 21 days or per physician order.

DETAILED DESCRIPTION:
Gaido Health's Remote Patient Monitoring Solution v1.0 is a wireless remote monitoring system intended for use by healthcare professionals for the collection of physiological data in home and healthcare settings. Patient information is displayed on a computer located at the medical institution. Every 15 minutes, a measurement is plotted on the User Interface of heart rate / respiration rate (by a Biovotion device). A non-invasive blood pressure (by an Omron device) along with an oral digital thermometer reading are taken per clinician orders and displayed on the Gaido dashboard. Wearable data are transmitted wirelessly from the Biovotion sensor (heart rate and respiratory rate) to the patient's smart phone that relays data to a cloud-based server for storage and analysis. Oral temperature and blood pressure are entered by the patient or care-giver into the patient's smart phone that relays data to a cloud-based server for storage.

The Remote Patient Monitoring system uses algorithms that indicate when patient vitals and patient reported outcomes have changed. Automatic patient surveys are sent to the patient with results displayed both on the computer located in the medical institution and the patient's smart phone. The patient surveys gather patient reported symptoms which are intended to be used in combination with vital signs to support decision-making. The system is intended for use with patients 18 years of age and older who are cared for by healthcare professionals.

ELIGIBILITY:
Inclusion Criteria:

1. Adult oncology patients over the age of 18 who are receiving chemotherapy.
2. Adult oncology in-patients over the age of 18 who are being being discharged.
3. Patients who have the mental capacity to understand how to use the devices and phone App; or patients who have a 24-hour caregiver who can manage the devices and complete patient surveys.
4. Patients who speak, read, and understand English.
5. Patients who have access to a smart phone.

Exclusion Criteria:

1. Non-English speaking patients.
2. Pregnant women.
3. Tattoos on outer side of upper arm (where the heart rate device will be worn).
4. Infant or pediatric (age less than 18).
5. Dementia, unless accompanied by a full-time caregiver.
6. Physically unable to wear the associated wearable devices; for example, amputees (preventing the placement of wearable devices worn on the arm).
7. Existence of open wounds or skin breakdown in the designated area for wearable device placement or on patients with conditions of irritable skin, per clinician judgment based on patient assessment.
8. Body mass index (BMI) >35 kg/m2, with conical shaped upper arms with significant adipose tissue (BP measurements might not perform properly).
9. Hospice patients who have an 'advanced directive'.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2019-09-09 (Estimated); Primary Completion 2019-11-30 (Estimated); Study Completion 2019-12-31 (Estimated)

PRIMARY OUTCOMES:
Feasibility of Gaido intervention for use by cancer patients | Evaluation last for 3 days after each patient use
  Feasibility will be measured through utilization of the intervention to track statistics such as wear time, completion of patient reported outcomes patients who are meet the criteria and are enrolled in the study. o Analysis of patient wear time for Gaido, using reporting tools as part of the Gaido solution.
  * Proportion of time that patients wear the Gaido solution
  * Proportion of participants completing self-reported symptom monitoring through the device
  * Proportion of participants completing vital sign data entry (blood pressure and oral temperature) through the device

SECONDARY OUTCOMES:
Acceptability of Gaido intervention for use by cancer patients | Evaluation last for 3 days after each patient use
  The research team will conduct semi-structured interviews with patients, to obtain feedback on usability and utility of the Gaido solution.
Potential impact of Gaido intervention on cancer patient outcomes | Evaluation last for 3 days after each patient use
  To describe health care utilization, potential conditions detected on patients receiving Remote Electronic Patient Monitoring.corresponding interventions on patients receiving Remote Electronic Patient Monitoring.The Electronic Health Record (EHR) will be used to validate the potential Gaido conditions/findings. The following information will be gathered from the EHR: clinical factors (e.g. activities of daily living, tumor staging, diagnosis dates, cancer treatment, prior cancer history, medical comorbidities, and current medications), health care utilization (e.g. inpatient admissions and emergency department visits), and end-of-life care (e.g. death date, hospice enrollment, location of death).

CONTACTS AND LOCATIONS:
Overall Officials: Philip Lowry, MD, Principal Investigator — Guthrie Medical Center
Locations (1):
- Guthrie Medical Center, Sayre, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No